CLINICAL TRIAL: NCT01737593
Title: Can Acetaminophen PO Given 1-2 Hours Before Bilateral Myringotomy Tube (BMT) Placement Reduce Emergence Agitation (EA) in Children After General Sevoflurane Anesthesia?
Brief Title: Can Acetaminophen Given 1-2 Hours to Children Before Ear Tube Surgery Reduce Agitation After Anesthesia?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis revealed a negative effect.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Wendy Ren, Physician, Assistant Clinical Professor-Pediatric Anesthesiology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 12-001510
Record Dates: First submitted 2012-11-13; First posted 2012-11-29 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-08

CONDITIONS: Emergence Agitation; Pain
Keywords: acetaminophen; emergence agitation; children; sevoflurane
MeSH Terms: conditions — Emergence Delirium; Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acetaminophen PR (Active Comparator): Acetaminophen PR (20-40mg/kg) after induction of Anesthesia (acetaminophen is in suppository form and given rectally)
  Interventions: Drug: Acetaminophen
- Acetaminophen PO-low dose (Active Comparator): Acetaminophen PO (10mg/kg) 60-120min before start of BMT placement (acetaminophen is in syrup form and given by mouth)
  Interventions: Drug: Acetaminophen
- Acetaminophen PO-high dose (Active Comparator): Acetaminophen PO (20mg/kg) 60-120min before start of BMT placement (acetaminophen is in syrup form and given by mouth)
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen
  Other Names: Tylenol

SUMMARY:
Emergence agitation (EA) occurs in up to 67% of pediatric patients after anesthesia for bilateral myringotomy tubes (BMT, "ear tubes"). The goal of this study is to find out whether acetaminophen given well before surgery can decrease pain and therefore, decrease emergence agitation better than acetaminophen given shortly before or during surgery. EA can be dangerous for the patient because it may be hard to monitor their vital signs during an important phase of recovery, they may injure themselves, may require the presence of extra staff, and it can be very distressing to the parents. Causes of EA are not well understood, but it can be worsened by pain. 70% of patients undergoing BMT experience pain that needs treatment. Intranasal fentanyl, a strong analgesic, has been shown to decrease EA, but often ends up in dose-dependent nausea and vomiting. In previous studies and in common practice, acetaminophen is given either 30 minutes before induction of anesthesia or immediately after induction. The peak analgesic effect of acetaminophen is 60-120 minutes. Since the procedure is generally completed in 5-10 minutes, the therapeutic effect of acetaminophen may not be present upon emergence from anesthesia.

The purpose of this study is to find out if acetaminophen given 60-120 minutes prior to emergence can decrease EA in patients undergoing BMT. Patients would be randomized to one of three groups: Control will receive acetaminophen rectally while under anesthesia (standard practice), Group 1 will receive acetaminophen 10 mg/kg at 60-120 minutes prior to surgery, Group 2 will receive acetaminophen 20 mg/kg at 60-120 minutes prior to surgery. All groups would also receive a dose of intranasal fentanyl during the surgery, which is standard practice. Patients would be observed in the recovery room at various time points for evidence of EA and pain.

DETAILED DESCRIPTION:
Emergence agitation (EA) occurs in up to 67% of patients undergoing Sevoflurane anesthesia for bilateral myringotomy tube placement (BMT). Often EA presents as inconsolable screaming, crying, thrashing, and kicking, and may require restraints. It can be dangerous for the patient because it may be difficult to monitor their vital signs during a critical phase of recovery (i.e. unable to detect hypoxemia), they may injure themselves as they thrash about, it usually requires the presence of extra staff, and it can be very distressing to the parents. Causes of EA are theoretical, but can be exacerbated by pain. 70% of patients undergoing BMT have pain requiring treatment. Since BMT is performed without IV placement the options for analgesia are limited to intranasal fentanyl, intramuscular ketorolac, rectal or oral acetaminophen, oral opioids (i.e. codeine, oxycodone). Intranasal Fentanyl has been shown to decrease EA, but results in post operative nausea and vomiting, as with any opioids. Intramuscular ketorolac is costly and can lead to hematomas. In previous studies (common practice), acetaminophen is given either 30 minutes before induction (PO route) or immediately after induction (PR route). Since the procedure is generally completed in 5-10 minutes, the therapeutic effect of acetaminophen can not be appreciated. The peak effect (for analgesia) of acetaminophen is 60-120 minutes. Our hypothesis: If acetaminophen is given 60-120 minutes prior to emergence, when it reaches therapeutic effect, it can decrease EA in patients undergoing BMT. The importance of mitigating EA not only involves patient safety and satisfaction, but will also impact hospital/surgery center efficiency (RN staffing and smoother and shorter recovery periods).

This study will be a randomized controlled trial. Potential subjects will be identified and recruited by study personnel and/or patient's surgeon. Children scheduled for BMT placement whose parents' consent to participate will be enrolled in the study. These patients will be consented on the day of surgery. Parents will be informed that whether they enroll their children in the study or not, they will be receiving standard clinical care. Only subjects meeting all inclusion criteria and requirements for continuation in the study will be consented.

Patients will be enrolled into one of three study groups. All patients meeting all inclusion criteria and requirements for the study (see below) will be identified, consented then computer randomized into either control, group 1 or 2.

Control - acetaminophen PR (20-40mg/kg) after induction of Anesthesia (acetaminophen is in suppository form and given rectally) Group 1 - acetaminophen PO (10mg/kg) 60-120min before start of BMT placement (acetaminophen is in syrup form and given by mouth) Group 2 - acetaminophen PO (20mg/kg) 60-120min before start of BMT placement (acetaminophen is in syrup form and given by mouth)

After randomization, treating physicians will be made aware of what treatment group the patient is assigned to. The data collection and behavior/pain assessments will be made by blinded study personnel in the operating room (only for induction) and PACU.

Data Collection: Data will be collected at the time points: Induction, Emergence (spontaneous extremity movement), and every 5 minutes after emergence until the patient is discharged. There will also be a follow-up questionnaire for the parent on satisfaction with the child's emergence, side effects, additional medications, and his/her PACU experience. This will be conducted on the phone within 36 hours after the parents have left the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients' ≥ 6 months - 6 years
* Patients must meet criteria for American Society of Anesthesiologists (ASA) physical status I, II.
* Patients must not be pre-medicated.
* Parents must give written consent on the surgery day and be able to sign informed consent form on the surgery day.
* Undergoing BMT surgery only.

Exclusion Criteria:

* Patients' <6 months and >6 years.
* Patients with known allergies to any of the medications used in this study.
* Patients with ASA status III & IV.
* Patients taking prescription pain medications prior to surgery.
* Patients taking medication that can cause drowsiness or alter mental status (eg. benzodiazepines, cough suppressants, diphenhydramine)
* Patients with significant history of psychiatric illness, neurologic disease (seizure disorder requiring medication therapy), and developmental delay.
* Patients have been pre-medicated.
* Patients undergoing other procedures that would prolong anesthetic exposure or confound post-operative pain.
* Intra-op complication that would require prolonged anesthetic exposure.
* If patient took acetaminophen prior to surgery and was not supposed to do so
* Patients that received ketorolac or additional analgesia during surgery.
* Patients that have liver disease.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Ren, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetaminophen PR: Acetaminophen PR (20-40mg/kg) after induction of Anesthesia (acetaminophen is in suppository form and given rectally)
  Acetaminophen
- Acetaminophen PO-low Dose: Acetaminophen PO (10mg/kg) 60-120min before start of BMT placement (acetaminophen is in syrup form and given by mouth)
  Acetaminophen
- Acetaminophen PO-high Dose: Acetaminophen PO (20mg/kg) 60-120min before start of BMT placement (acetaminophen is in syrup form and given by mouth)
  Acetaminophen
Period: Overall Study
Arm/Group | Acetaminophen PR | Acetaminophen PO-low Dose | Acetaminophen PO-high Dose
Started | 37 | 32 | 39
Completed | 37 | 32 | 39
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen PR | Acetaminophen PO-low Dose | Acetaminophen PO-high Dose | Total
Number analyzed (Participants) | 37 | 32 | 39 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.08 (1.39) | 2.20 (1.58) | 2.31 (1.53) | 2.23 (1.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 17 | 37
  Male | 29 | 20 | 22 | 71
Region of Enrollment [Number; unit: participants]
  United States | 37 | 32 | 39 | 108

OUTCOME MEASURES:

1. Primary Outcome: Postanesthesia Emergence Agitation (EA) Score
Description: EA was evaluated using the Pediatric Anesthesia Emergence Delirium (PAED) scale. This scale measures if the: 1. Child makes eye contact with the caregiver, 2. Child's actions are purposeful, 3. Child is aware of his/her surroundings, 4. Child is restless, 5. Child is inconsolable.
  Items 1, 2, and 3 are reversed scored as follows: 4 _ not at all, 3 _ just a little, 2 _ quite a bit, 1 _ very much, 0 _ extremely. Items 4 and 5 are scored as follows: 0 _ not at all, 1 _ just a little, 2 _ quite a bit, 3 _ very much, 4_extremely. Scores of each item are summed to obtain a total PAED scale score, range 0-20, with higher PAED scores indicating a greater degree of emergence delirium.
  The average PAED score of all the time points is use
Time Frame: Induction,Emergence(spontaneous extremity movement),and every 5 min after emergence until the patient is discharged. This is an average of 3 hours till discharge.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Acetaminophen by Rectum (PR): Acetaminophen PR (20-40mg/kg) after induction of Anesthesia (acetaminophen is in suppository form and given rectally)
  Acetaminophen
- Acetaminophen by Mouth (PO) - Low Dose: Acetaminophen PO (10mg/kg) 60-120min before start of BMT placement (acetaminophen is in syrup form and given by mouth)
  Acetaminophen
- Acetaminophen by Mouth (PO) - High Dose: Acetaminophen PO (20mg/kg) 60-120min before start of BMT placement (acetaminophen is in syrup form and given by mouth)
  Acetaminophen
Arm/Group | Acetaminophen by Rectum (PR) | Acetaminophen by Mouth (PO) - Low Dose | Acetaminophen by Mouth (PO) - High Dose
Number analyzed (Participants) | 37 | 32 | 39
units on a scale | 5.63 (3.07) | 6.19 (3.53) | 6.37 (3.96)

2. Secondary Outcome: Postanesthesia Pain Score
Description: Children's Hospital of Eastern Ontario pain scale (CHEOPS) is an observational scale for measuring postoperative pain in young children. The scale includes six categories of pain behavior: (Cry, facial, verbal, torso, touch, and legs). A score ranging from 0 to 2 or 1 to 3 is assigned to each activity and the summed score ranges between 4 and 13, with a higher score meaning more pain.
Time Frame: Induction
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Acetaminophen PO - Low Dose: Acetaminophen PO (10mg/kg) 60-120min before start of BMT placement (acetaminophen is in syrup form and given by mouth)
  Acetaminophen
- Acetaminophen PO - High Dose: Acetaminophen PO (20mg/kg) 60-120min before start of BMT placement (acetaminophen is in syrup form and given by mouth)
  Acetaminophen
Arm/Group | Acetaminophen PR | Acetaminophen PO - Low Dose | Acetaminophen PO - High Dose
Number analyzed (Participants) | 37 | 32 | 39
units on a scale | 7.78 (1.931) | 8.66 (2.444) | 8.69 (2.307)

3. Secondary Outcome: Postanesthesia Pain Score
Description: as for outcome 2
Time Frame: Emergence (spontaneous extremity movement)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen PR | Acetaminophen PO - Low Dose | Acetaminophen PO - High Dose
Number analyzed (Participants) | 37 | 32 | 39
units on a scale | 9.0 (1.780) | 8.56 (1.564) | 8.79 (1.689)

4. Secondary Outcome: Postanesthesia Pain Score
Description: as for outcome 2
Time Frame: 5 minutes post-emergence
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen PR | Acetaminophen PO - Low Dose | Acetaminophen PO - High Dose
Number analyzed (Participants) | 37 | 32 | 39
units on a scale | 8.27 (2.244) | 8.41 (1.643) | 8.08 (2.044)

5. Secondary Outcome: Postanesthesia Pain Score
Description: as for outcome 2
Time Frame: 15 minutes post-emergence
Population: Participants not yet discharged at the 15 minute time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen PR | Acetaminophen PO - Low Dose | Acetaminophen PO - High Dose
Number analyzed (Participants) | 36 | 32 | 39
units on a scale | 6.83 (1.577) | 7.22 (1.518) | 7.36 (1.814)

6. Secondary Outcome: Postanesthesia Pain Score
Description: as for outcome 2
Time Frame: 30 minutes post-emergence
Population: Participants not yet discharged at the 30 minute time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen PR | Acetaminophen PO - Low Dose | Acetaminophen PO - High Dose
Number analyzed (Participants) | 33 | 27 | 33
units on a scale | 6.52 (1.278) | 6.78 (1.251) | 6.42 (1.458)

7. Secondary Outcome: Postanesthesia Pain Score
Description: as for outcome 2
Time Frame: 45 minutes post-emergence
Population: Participants not yet discharged at the 45 minute time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen PR | Acetaminophen PO - Low Dose | Acetaminophen PO - High Dose
Number analyzed (Participants) | 13 | 11 | 14
units on a scale | 6.77 (1.301) | 6.18 (0.751) | 6.71 (1.326)

8. Secondary Outcome: Postanesthesia Pain Score
Description: as for outcome 2
Time Frame: Prior to discharge, up to 3 hours after induction.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen PR | Acetaminophen PO - Low Dose | Acetaminophen PO - High Dose
Number analyzed (Participants) | 37 | 32 | 39
units on a scale | 5.95 (0.848) | 6.03 (0.999) | 5.92 (1.244)

ADVERSE EVENTS:
Arm/Group | Acetaminophen PR | Acetaminophen PO-low Dose | Acetaminophen PO-high Dose
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/32 | 0/39
Other Adverse Events (participants affected / at risk) | 0/37 | 0/32 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No